CLINICAL TRIAL: NCT00232375
Title: Intervention to Preserve Beta-Cell Function in GAD Ab-Positive Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-81
Record Dates: First submitted 2005-09-29; First posted 2005-10-04 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-01

CONDITIONS: GAD Ab Positive Clinically Type 2 Diabetic Patients
Keywords: SPIDDM; LADA; GAD antibody; Beta cell function; Insulin
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin

INTERVENTIONS:
Drug: Insulin

SUMMARY:
We tested the hypothesis that insulin therapy rather than sulfonylurea (SU) treatment has a preferable outcome to reverse or preserve beta cell function in the patients with diabetes that is called slowly progressive insulin-dependent (type 1) diabetes (SPIDDM) or latent autoimmune diabetes in adult (LADA).

DETAILED DESCRIPTION:
In a multicenter, randomized, nonblinded clinical study, 4,089 non-insulin dependent diabetic patients were screened for glutamic acid decarboxylase autoantibodies (GADAb). Sixty GADAb-positive non-insulin requiring diabetic patients with duration of diabetes =/<5 years were assigned to either the SU group (n = 30) or the Insulin group (n = 30). Serum C-peptide response to annual oral glucose tolerance tests were followed for 57 mean months. The primary endpoint was insulin-dependency (IDDM: integrated C-peptide values [sigma C-peptide] <4 ng/ml).

ELIGIBILITY:
Inclusion Criteria:

* Subjects should use SU agents to obtain as a goal good glycemic control.
* Duration of diabetes within 5 years from the onset (or diagnosis).

Exclusion Criteria:

* Subjects having history of hyperglycemia requiring insulin treatment and/or history of ketosis/ketoacidosis were excluded.
* Subjects with malignant diseases, systemic inflammatory diseases, renal or liver disorders or malabsorption were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 1996-01; Study Completion 2005-01

PRIMARY OUTCOMES:
The primary endpoint was insulin-dependency (IDDM: integrated C-peptide values [sigma C-peptide] <4 ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Tetsuro Kobayashi, Professor, Study Director — Third Department of Internal Medicine, Interdisciplinary Graduate School of Medicine and Engineering, University of Yamanashi
Locations (1):
- University of Yamanashi, Tamaho, Yamanashi, Japan

REFERENCES:
- [Derived] Maruyama T, Tanaka S, Shimada A, Funae O, Kasuga A, Kanatsuka A, Takei I, Yamada S, Harii N, Shimura H, Kobayashi T. Insulin intervention in slowly progressive insulin-dependent (type 1) diabetes mellitus. J Clin Endocrinol Metab. 2008 Jun;93(6):2115-21. doi: 10.1210/jc.2007-2267. Epub 2008 Apr 8. PMID 18397986